CLINICAL TRIAL: NCT05506423
Title: An Observational Registry Study of Safety and Effectiveness Outcomes Through 24 Months Postoperatively Following CycloPen™ Micro-Interventional Cyclodialysis System Procedures in Patients With Open Angle Glaucoma
Brief Title: Study of the CycloPen Micro-Interventional System and Long-Term Clinical Outcomes
Acronym: CREST
Status: Enrolling by invitation | Type: Observational
Sponsor: Iantrek, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ITR-CYC-041
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- CycloPen Cyclodialysis System in conjunction with cataract surgery: Ophthalmic surgical intervention with the CycloPen Cyclodialysis System in conjunction with cataract surgery
  Interventions: Device: CycloPen Cyclodialysis System
- CycloPen Cyclodialysis System in standalone surgery: Ophthalmic surgical intervention with the CycloPen Cyclodialysis System
  Interventions: Device: CycloPen Cyclodialysis System

INTERVENTIONS:
Device: CycloPen Cyclodialysis System — The CycloPen Micro-Interventional Cyclodialysis System is used to create and cyclodialysis cleft and deliver allograft scleral tissue and/or viscous material to reinforce and maintain the cleft postoperatively.

SUMMARY:
This observational study will enroll adults with open angle glaucoma (OAG) who had surgery to reduce intraocular pressure (IOP) using the CycloPen Micro-Interventional System. Consenting participants will be followed for 24 months after their surgery.

Data regarding IOP, use of glaucoma medications, and any side effects related to the surgery will be collected from participants' preoperative examination, their surgery, and postoperative examinations.

DETAILED DESCRIPTION:
This is a multicenter, observational registry of eligible adults with open angle glaucoma (OAG) in whom IOP-lowering surgery with the CycloPen Micro-Interventional System was performed are consecutively enrolled.

Data will be collected from the preoperative visit(s) that directly preceded surgery, the surgical procedure, and postoperative visits through 24 months after CycloPen System use.

Specific data to be collected includes details of the CycloPen surgical procedure, IOP, use of ocular hypotensive medications, and any side effects related to the surgery.

ELIGIBILITY:
To be included, participants must have:

1. Open angle glaucoma
2. IOP-lowering surgical procedure using the CycloPen System

There are no exclusionary criteria.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants who underwent IOP-lowering surgical procedures using the CycloPen Micro-Interventional System for uveoscleral outflow enhancement
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Percent of eyes with intraocular pressure (IOP) reduction ≥ 20% in comparison with baseline | 12 months postoperative
  Intraocular pressure (IOP) is at least 20% lower than before surgery without additional ocular hypotensive medications or IOP-lowering surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tsontcho Ianchulev, MD, Study Chair — Iantrek, Inc.
Locations (16):
- United States (15):
  - CREST Site 05, Newport Beach, California
  - CREST Site 03, Cape Coral, Florida
  - CREST Site 10, DeLand, Florida
  - CREST Site 06, Fort Myers, Florida
  - CREST Site 07, Atlanta, Georgia
  - CREST Site 12, Chevy Chase, Maryland
  - CREST Site 13, Rockville, Maryland
  - CREST Site 16, Las Vegas, Nevada
  - CREST Site 14, New Brunswick, New Jersey
  - CREST Site 15, New York, New York
  - CREST Site 17, Williamsville, New York
  - CREST Site 01, Fort Washington, Pennsylvania
  - CREST Site 04, Crossville, Tennessee
  - CREST Site 09, Fort Worth, Texas
  - CREST Site 11, Salt Lake City, Utah
- CREST Site 301, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barber K, Flowers B, Patterson M, Vera L, Ianchulev T, Ahmed II. Bio-interventional uveoscleral outflow enhancement in patients with medically uncontrolled primary open-angle glaucoma: 1-year results of allograft-reinforced cyclodialysis. Ther Adv Ophthalmol. 2025 Aug 11;17:25158414251362010. doi: 10.1177/25158414251362010. eCollection 2025 Jan-Dec. PMID 40799662